CLINICAL TRIAL: NCT03982615
Title: The Laser-Lok Trial: Impact of Laser-modified Abutment Topography on Peri-implant Mucosal Integration
Brief Title: Impact of Laser-modified Abutment Topography on Peri-implant Mucosal Integration
Acronym: Laser-Lok
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Lyndon F Cooper, Associate Dean of Research, Chair-Department of Oral Biology, College of Dentistry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1358
Record Dates: First submitted 2019-05-21; First posted 2019-06-11 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Dental Implant Failure Nos
Keywords: RNASeq; mucosal integration

STUDY DESIGN:
Intervention Model Description: Prospective randomized split mouth designed study intended to evaluate the healing and health of peri-implant mucosa following placement of titanium abutments with or without laser-etching.
  Each subject will receive two dental implants. One implant will receive (by randomization) a laser-etched ("Laser-Lok") abutment. The other implant will receive a standard healing abutment (not laser-etched).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laser-Lok abutment (Experimental): Laser-etched abutment
  Interventions: Device: Laser-Lok abutment
- Standard Healing abutment (Active Comparator): Standard abutment which is not laser-etched
  Interventions: Device: Standard healing abutment

INTERVENTIONS:
Device: Laser-Lok abutment — Each subject will receive two dental implants. One implant will receive (by randomization) a laser-etched ("Laser-Lok") abutment.
  Other Names: laser-etched abutment
  Arms: Laser-Lok abutment
Device: Standard healing abutment — Each subject will receive two dental implants. One implant will receive (by randomization) receive a standard healing abutment (not laser-etched).
  Other Names: non-laser etched abutment
  Arms: Standard Healing abutment

SUMMARY:
This study is a prospective randomized split mouth study intended to evaluate the healing and health of peri-implant mucosal tissue following placement of titanium abutments with or without laser-etching.

Each subject will receive two implants. Following placement of the two 4.2mm diameter implants, one implant will receive (by randomization) a laser-etched abutment ('Laser-Lok'). The other implant will receive a standard, non-etched healing abutment. Subjects will be sequentially subdivided into four groups (n=5) and scheduled for a biopsy of the peri-implant tissues of both implants at either 8 weeks, 4 weeks, 2 weeks or 1 week after implant surgery. These biopsies, about the size of a grain of rice, will be analyzed using immunohistochemical and RNASeq techniques to identify molecular changes in response to laser etching.

At approximately 8 weeks after implant surgery, subjects will have abutments removed from both implants and digital impressions taken for final crown fabrication. At approximately 11-12 weeks after implant surgery, final crowns will be placed. Subjects return to clinic at approximately 1 year post surgery for a final study visit to assess the peri-implant mucosa surrounding both implants as measured by bleeding upon probing, probing depth and peri-apical radiography.

DETAILED DESCRIPTION:
A dental implant is an artificial "root" for a missing tooth made out of surgical grade metals, usually titanium, which is placed in the jaw. An implant is designed to provide a strong foundation for an artificial replacement tooth, also called a "crown". An abutment is a medical grade connector, usually made of titanium, which is placed on top of the implant, and is designed to hold and connect the crown to the implant. A crown, also called a "dental cap" is an artificial tooth, generally made of porcelain or surgical grade metals.

Osseointegration is defined as the fusion of a dental implant and abutment with the surrounding jaw bone and is a critical step during implant therapy. During this process, the titanium and bone need to become one solid structure (without any intervening inflammatory mucosal tissue in between) for optimum strength and viability.

It is hypothesized that use of an abutment whose surface has been etched with a laser ("laser-etched") will enhance the attachment of the abutment to the surrounding bone and mucosal tissue and optimize healing.

The goal of this research is to compare, by split mouth design, the healing process of peri-implant mucosal tissue adjacent to a standard healing abutment (not laser-etched) versus mucosal tissue healing adjacent to a laser-etched abutment .

Each subject will receive two implants. One implant will receive (by randomization) a standard titanium healing abutment that is not laser-etched. The other implant will receive a laser-etched ("Laser-Lok") abutment. Subjects will be sequentially subdivided into 4 groups (n=5) and scheduled for a biopsy of peri-implant tissue at both implant sites at either 8 weeks, 4 weeks, 2 weeks or 1 week after implant surgery. The biopsies, about the size of a grain of rice, will be analyzed using histological and molecular techniques to identify cellular changes in response to laser-etching.

Approximately 8 weeks after implant placement, subject will have abutments removed and digital impressions taken for final crown fabrication. At approximately 11-12 weeks post implant placement, final crowns will be placed. Subjects return to clinic at approximately 1 year post surgery for a final study visit to assess the peri-implant mucosa around both implants as measured by bleeding upon probing, probing depth and peri-apical radiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult, able to provide informed written consent and available for 1 year follow-up visit
* Have 2 edentulous sites requiring single tooth implants for restoration in two separate quadrants
* Implant sites must be restorable with 4.2mm diameter implants
* Have natural teeth adjacent (at least unilaterally) to proposed implant sites
* Able to pay for implant crowns at UIC College of Dentistry postgraduate fees to complete treatment

Exclusion Criteria:

* Uncontrolled/rampant caries or periodontal disease
* Unable to demonstrate adequate home oral hygiene
* smoker within the past 6 months
* ASA Class 3+, immune-compromised
* Pregnant or planning to become pregnant within 6 months
* Severe bruxism
* History of bisphosphonate use
* Bone grafting required for implant placement
* Missing tooth is too small to be restored using a 4.2mm implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Molecular profiling of peri-implant mucosal tissues | 1 week, 2 week, 4 week, and 8 week after implant surgery
  Fold change (> 2 fold) expression of junctional epithelial gene expression (e.g. ODAM., FDSCP)

SECONDARY OUTCOMES:
Radiographic parameter | 1 week and 1 year post implant surgery
  mm change (> 0.1 mm) in peri-implant bone levels at mesial and distal positions

OTHER OUTCOMES:
Peri-implant probing depth | 1 week and 1 year post implant surgery
  in mm
Bleeding on probing | 1 week and 1 year post implant surgery
  yes/no at mesial, distal, buccal and lingual positions
Gingival Index | 1 week and 1 year post implant surgery
  tissue redness 1 - 4

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon F Cooper, DDS, PhD, Principal Investigator — University of Illinois at Chicago College of Dentistry
Locations (1):
- University of Illinois at Chicago, College of Dentistry, Clinical Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leong A, De Kok I, Mendonca D, Cooper LF. Molecular Assessment of Human Peri-implant Mucosal Healing at Laser-Modified and Machined Titanium Abutments. Int J Oral Maxillofac Implants. 2018 Jul/Aug;33(4):895-904. doi: 10.11607/jomi.6367. PMID 30025007